CLINICAL TRIAL: NCT02079805
Title: A Study to Explore the Effects of Azilsartan Compared to Telmisartan on Insulin Resistance of Patients With Essential Hypertension on Type 2 Diabetes Mellitus by HOMA-R
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 279/NRP-001; U1111-1151-7168 (Registry Identifier: UTN (WHO)); AZI-P4-004 (Other: Takeda); JapicCTI-142461 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Essential Hypertension Complicated by Type 2 Diabetes Mellitus
MeSH Terms: interventions — azilsartan; Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azilsartan 20 mg (Experimental): Participants will receive azilsartan 20 mg once daily in the morning before or after breakfast.
  Interventions: Drug: Azilsartan
- Telmisartan 40 mg (Active Comparator): Participants will receive telmisartan 40 mg once daily in the morning before or after breakfast.
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Azilsartan — Azilsartan tablets
  Other Names: Azilva Tablets
  Arms: Azilsartan 20 mg
Drug: Telmisartan — Telmisartan tablets
  Other Names: Micardis Tablets
  Arms: Telmisartan 40 mg

SUMMARY:
Multicenter, randomized, open-label, parallel-group exploratory study to explore the effects of azilsartan (Azirva), compared with telmisartan, on insulin resistance in participants with essential hypertension complicated by type 2 diabetes mellitus

DETAILED DESCRIPTION:
The primary objective of the present study is to explore the effects of azilsartan 20 mg, compared with telmisartan 40 mg, once daily orally for 12 weeks on insulin resistance in participants with essential hypertension complicated by type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. The participant was given the diagnosis of grade I or II essential hypertension and was judged by the principal investigator or investigator that they can be appropriately treated with azilsartan 20 mg and telmisartan 40 mg.
2. Sitting systolic blood pressure of ≥ 130 mmHg and < 180 mmHg or sitting diastolic blood pressure of ≥ 80 mmHg and < 110 mmHg at the start of the treatment period (Week 0) Sitting blood pressure will be measured until 2 consecutive stable measurements are obtained (i.e., the difference between 2 measurements: diastolic blood pressure of <5 mmHg and systolic blood pressure of < 10 mmHg) after resting in a sitting position for at least 5 minutes. The average value of the last 2 measurements will be recorded (the first the decimal place is rounded off).
3. Type 2 diabetes mellitus
4. HbA1c (NGSP (National Glycohemoglobin Standardization Program) value) of < 8.4% during 3 months before informed consent, with a ≤ 0.3% change in HbA1c (peak minus nadir) during 3 months before informed consent
5. No change in diet/exercise therapy during the 3 months before the informed consent in a participant who has been on diet/exercise therapy and instructed to improve life style (e.g., diet and exercise)
6. Age ≥ 20 years at the time of consent
7. Outpatients
8. Capable of providing written consent before participation in this study.

Exclusion Criteria:

1. Grade III essential hypertension (i.e., sitting systolic blood pressure 180 mmHg or sitting diastolic blood pressure ≥ 110 mmHg), secondary hypertension, or malignant hypertension.
2. Grade II essential hypertension (i.e., sitting systolic blood pressure ≥ 160 mmHg or sitting diastolic blood pressure ≥ 100 mmHg) for which antihypertensive drug(s) are used
3. Use of oral antihypertensive medication within 2 weeks before the start of the treatment period Participants who are on any antihypertensive agent at the time of informed consent can be enrolled in the study only after 2-week washout following informed consent.
4. Use of RAS inhibitors or thiazolidines within 3 months before the start of the treatment period
5. Type 1 diabetes mellitus
6. Fasting blood glucose of < 180 mg/dL and HOMA-R of ≤ 1.6 at the start of the treatment period (Week 0)
7. Receiving or requiring any of the following at the time of informed consent:

   * Insulin, glucagon-like peptide-1 (GLP-1) receptor agonists, or other parenteral hypoglycemic agents
   * Combination therapy with 3 or more oral hypoglycemic agents
8. Change of antidiabetic medication (including dosage change) within 3 months before the start of the treatment period
9. Having diagnosed/treated any of the following cardiovascular diseases within 3 months before the start of the treatment period:

   * Cardiac disease/condition: myocardial infarction, coronary revascularization procedure
   * Cerebrovascular disease: cerebral infarction, cerebral haemorrhage, transient ischaemic attack
   * Advanced hypertensive retinopathy (retinal bleeding or oozing, papilloedema)
10. Having diagnosed/treated for any of the following cardiovascular diseases more than 3 months before the start of the treatment period, and is now still in unstable condition.

    * Cardiac disease/condition: myocardial infarction, coronary revascularization procedure
    * Cerebrovascular disease: cerebral infarction, cerebral haemorrhage, transient ischaemic attack
11. Past or current history of any of the following cardiovascular diseases.

    * Cardiac valve stenosis
    * Angina pectoris requiring medication
    * Congestive cardiac failure requiring medication
    * Arrhythmia requiring medication (e.g., paroxysmal atrial fibrillation, severe bradycardia, torsade de pointes, and ventricular fibrillation)
    * Arteriosclerosis obliterans with intermittent claudication or other symptoms
12. Have severe ketosis, diabetic coma or precoma, severe infection, or serious trauma
13. Clinically evident renal disorder (e.g., eGFR <30 mL/min/1.73 m2)
14. Markedly low bile secretion or severe hepatic disorder
15. History of hypersensitivity or allergy to azilsartan or telmisartan or to both.
16. Presence of hyperkalemia (potassium level ≥ 5.5 mEq/L on laboratory testing)
17. Currently participating in any other clinical study.
18. Pregnant women, women with possible pregnancy, or breast-feeding women.
19. Other participants who are inappropriate for participation in this study in the opinion of the principal investigator or investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda
Locations (1):
- Kyoto, Kyoto, Japan

REFERENCES:
- [Derived] Naruse M, Koike Y, Kamei N, Sakamoto R, Yambe Y, Arimitsu M. Effects of azilsartan compared with telmisartan on insulin resistance in patients with essential hypertension and type 2 diabetes mellitus: An open-label, randomized clinical trial. PLoS One. 2019 Apr 3;14(4):e0214727. doi: 10.1371/journal.pone.0214727. eCollection 2019. PMID 30943275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 27 investigative sites in Japan, from 04 June 2014 to 25 April 2016.
Pre-assignment Details: Participants with diagnosis of type 2 diabetes mellitus were enrolled in 2 treatment group: Azilsartan 20 mg, and Telmisartan 40 mg for 12 weeks as treatment period.
Groups:
- Telmisartan 40 mg: Participants received telmisartan 40 mg, once daily in the morning before or after breakfast for 12 weeks as treatment priod.
- Azilsartan 20 mg: Participants received azilsartan 20 mg, once daily in the morning before or after breakfast for 12 weeks as treatment priod.
Period: Overall Study
Arm/Group | Telmisartan 40 mg | Azilsartan 20 mg
Started | 16 | 17
Completed | 16 | 15
Not Completed | 0 | 2
Not completed — Pretreatment Event/Adverse Event | 0 | 1
Not completed — Voluntary Withdrawal | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan 40 mg | Azilsartan 20 mg | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (9.10) | 63.2 (12.76) | 64.2 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 7 | 7 | 14
Weight [Mean (Standard Deviation); unit: kg] | 70.95 (16.689) | 70.41 (14.878) | 70.67 (15.534)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 27.18 (3.720) | 27.19 (4.642) | 27.19 (4.154)
Smoking Classification [Number; unit: participants]
  Never smoked | 8 | 8 | 16
  Current smoker | 2 | 3 | 5
  Ex-smoker | 6 | 6 | 12
Alcohol Classification [Number; unit: participants] — Participants who answered Yes or No for a question "Drik Alcohol Almost Everyday?" were reported.
  participants
    Yes | 6 | 5 | 11
    No | 10 | 12 | 22
Duration of Hypertention [Mean (Standard Deviation); unit: Years] | 4.71 (4.391) | 3.54 (4.392) | 4.11 (4.363)
Duration of Diabetes Mellitus [Mean (Standard Deviation); unit: Years] | 4.53 (4.279) | 4.89 (5.039) | 4.72 (4.617)
Taking Biguanides [Number; unit: participants] — Participants who had taken biguanides when study started were reported.
  participants
    Had taken | 3 | 4 | 7
    Not had taken | 13 | 13 | 26
Insulin Resistance Index (HOMA-R) [Mean (Standard Deviation); unit: HOMA-R Score] — Insulin Resistance Index (HOMA-R) measures insulin resistance, calculated by fasting insulin (μU/mL) multiplied by fasting glucose (mg/dL), and divided by a constant (405). A higher score indicates higher insulin resistance.
  HOMA-R Score | 3.31 (1.366) | 4.24 (1.843) | 3.79 (1.671)
Blood Pressure Systolic Mean [Mean (Standard Deviation); unit: mmHg] | 145.6 (9.91) | 143.3 (9.28) | 144.4 (9.51)
Blood Pressure Diastolic Mean [Mean (Standard Deviation); unit: mmHg] | 89.3 (10.61) | 88.8 (7.19) | 89.0 (8.87)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent] — Glycosylated Hemoglobin (HbA1c) were caluculated by the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound.
  percent | 6.63 (0.411) | 6.81 (0.488) | 6.72 (0.454)

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Resistance Index (HOMA-R) From Baseline at the End of the Treatment Period (Week 12)
Description: Change from the start of the treatment period (baseline) at the end of the treatment period (Week 12) was reported. Insulin Resistance Index (HOMA-R) measures insulin resistance, calculated by fasting insulin (μU/mL) multiplied by fasting glucose (mg/dL), and divided by a constant (405).
Time Frame: Baseline and Week 12
Population: The full analysis set was defined as the participants who received at least 1 dose of the study drug for the treatment period.
Measure: Mean (Standard Deviation); unit: HOMA-R Score
Arm/Group | Telmisartan 40 mg | Azilsartan 20 mg
Number analyzed (Participants) | 16 | 16
HOMA-R Score | -0.23 (0.928) | 0.22 (2.449)
Statistical Analysis 1: Comparison: Telmisartan 40 mg vs Azilsartan 20 mg; Telmisartan 40 mg, Azilsartan 20 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.44, 95% CI 2-sided [-0.89 to 1.78]

2. Secondary Outcome: Change in Fasting Blood Glucose From Baseline at the End of the Treatment Period (Week 12)
Description: Change from baseline in fasting blood glucose values collected at week 12 or final visit relative to baseline was reported.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Telmisartan 40 mg | Azilsartan 20 mg
Number analyzed (Participants) | 16 | 16
mg/dL | -1.06 (14.991) | 2.00 (18.308)

3. Secondary Outcome: Change in Fasting Insulin From Baseline at the End of the Treatment Period (Week 12)
Description: Change from baseline in fasting insulin values collected at week 12 or final visit relative to baseline was reported.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µU/mL
Arm/Group | Telmisartan 40 mg | Azilsartan 20 mg
Number analyzed (Participants) | 16 | 16
µU/mL | -0.818 (2.7623) | 0.475 (6.3847)

4. Secondary Outcome: Change in Glycosylated Hemoglobin (HbA1c) From Baseline at the End of the Treatment Period (Week 12)
Description: Change from baseline in the values of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 or final visit relative to baseline was reported.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Telmisartan 40 mg | Azilsartan 20 mg
Number analyzed (Participants) | 16 | 17
percent | 0.10 (0.290) | 0.09 (0.382)

5. Secondary Outcome: Change in Homeostasis Model Assessment of Beta Cell Function (HOMA-β) From Baseline at the End of the Treatment Period (Week 12)
Description: Change from baseline in HOMA-β collected at week 12 or final visit relative to baseline was reported. Homeostasis model assessment of beta cell function measures as following; HOMA-β = fasting insulin (μU/mL) ×360/{fasting glucose (mg/dL) - 63}.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Telmisartan 40 mg | Azilsartan 20 mg
Number analyzed (Participants) | 16 | 16
percent | -3.88 (20.151) | -0.44 (30.985)

6. Secondary Outcome: Change in 1,5-anhydroglucitol (1,5-AG) From Baseline at the End of the Treatment Period (Week 12)
Description: Change from baseline in 1,5-G concentration collected at week 12 or final visit relative to baseline was reported.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Telmisartan 40 mg | Azilsartan 20 mg
Number analyzed (Participants) | 16 | 16
μg/mL | 0.24 (2.143) | -0.66 (2.454)

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Time Frame: Up to Week 12
Population: The safety analysis set was defined as the participants who received at least 1 dose of the study drug for the treatment period.
Measure: Number; unit: participants
Arm/Group | Telmisartan 40 mg | Azilsartan 20 mg
Number analyzed (Participants) | 16 | 17
participants | 8 | 6

ADVERSE EVENTS:
Time Frame: Up to Week 12
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Telmisartan 40 mg | Azilsartan 20 mg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 8/16 | 6/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 40 mg (N=16) | Azilsartan 20 mg (N=17)
Diabetic retinopathy (Eye disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Blood pressure decreased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cutaneous amyloidosis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.